CLINICAL TRIAL: NCT01069133
Title: Effect of Rifaximin Therapy on Brain Activation in Patients With Minimal Hepatic Encephalopathy Using Functional MR, MR Spectroscopy,Diffusion Tensor Imaging Microbiome and Metabolome: a Prospective Trial
Brief Title: Study of Rifaximin in Minimal Hepatic Encephalopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Jasmohan Bajaj, Associate Professor of Medicine, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAJAJ010
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Minimal Hepatic Encephalopathy
Keywords: minimal hepatic encephalopathy; cirrhosis; complications
MeSH Terms: conditions — Fibrosis | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rifaximin (Experimental)
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — 550mg BID open-label
  Other Names: xifaxan
Drug: rifaximin — 550mg PO BID
  Other Names: xifaxan

SUMMARY:
Rifaximin therapy will improve brain functioning on MRI scanning and change the microbiome and metabolome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* cirrhosis diagnosed by clinical or biopsy grounds
* Minimal hepatic encephalopathy defined by impaired performance on at least 2 of the following: number connection tests A/B, digit symbol and block design tests (NCT-A, NCT-B, DST and BDT) compared to age and education-matched controls.
* No contraindications to MRI
* TIPS (transjugular intra-hepatic porto-systemic shunt) procedure or elective surgery planned within the next 8 weeks

Exclusion Criteria:

* Current therapy with lactulose, rifaximin or other treatment for hepatic encephalopathy.
* Prior episodes of overt HE
* MMSE <25
* TIPS placement
* Unable to give informed consent.
* Contra-indications to MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
brain activation on fMRI | 2 months
Microbiome constituents | 8 weeks

SECONDARY OUTCOMES:
brain edema and brain metabolite concentration | 2 months
Metabolome of urine and serum | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, MSc, Principal Investigator — McGuire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

REFERENCES:
- [Derived] Bajaj JS, Heuman DM, Sanyal AJ, Hylemon PB, Sterling RK, Stravitz RT, Fuchs M, Ridlon JM, Daita K, Monteith P, Noble NA, White MB, Fisher A, Sikaroodi M, Rangwala H, Gillevet PM. Modulation of the metabiome by rifaximin in patients with cirrhosis and minimal hepatic encephalopathy. PLoS One. 2013;8(4):e60042. doi: 10.1371/journal.pone.0060042. Epub 2013 Apr 2. PMID 23565181